CLINICAL TRIAL: NCT02201875
Title: Study of Periodic Breathing in Healthy Humans
Brief Title: Intrinsic Periodic Pattern of Breathing
Acronym: PERHYP1
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Association pour la Recherche en Physiologie de l'Environnement (Other)
Responsible Party: Principal Investigator, Pr. Jean Paul RICHALET, Director of Department, Association pour la Recherche en Physiologie de l'Environnement
Other Study IDs: PERHYP1
Record Dates: First submitted 2014-01-22; First posted 2014-07-28 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-07

CONDITIONS: Normoxia; Hypoxia; Hyperoxia; Hypercapnia
Keywords: hypoxia; exercise; periodic breathing; hypercapnia; apneas; cardiac failure
MeSH Terms: conditions — Hypoxia; Hyperoxia; Hypercapnia; Motor Activity; Apnea; Heart Failure

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Healthy subjects: male, aged 18-65 moderately trained healthy, no treatment
- obstructive sleep apneas: patients with apnea/hypopnea index > 15 BMI < 30 Age < 50 yrs
- cardiac failure: NYHA class I to III ejection fraction < 40% age < 65 yrs BMI < 30

SUMMARY:
We made a fortuitous observation of periodic breathing in a healthy subject coming to our outpatient mountain medicine consultation at Avicenne hospital in Bobigny (France). During this consultation, subjects perform a hypoxia exercise test, which allows a good prediction of their risk factors for severe high altitude illnesses. Surprisingly, breath-by-breath recording of the ventilation signal showed a periodic breathing pattern, which increased when the subject started to exercise in hypoxic conditions and was maintained during normoxic exercise.

Therefore, our objective was to confirm this observation in a retrospective study led in 82 subjects who passed this test. We tested the hypothesis that subjects with a brisk ventilatory response to hypoxia might show a more pronounced periodic pattern of ventilation, due to a higher gain of the chemoreceptor feedback loop. Then, our objective is to investigate the mechanisms involved in the periodic pattern in healthy subjects, as a function of exercise intensity, altitude intensity, role of peripheral and central chemoreceptors to O2 and CO2. Finally, we want to investigate the possible role of this ventilatory instability in patients with obstructive or central apneas.

DETAILED DESCRIPTION:
In a preliminary study, among the population coming to the outpatient consultation of mountain medicine at Avicenne hospital in 2012, 82 subjects (38 females and 44 males) were randomly selected and separated in two groups of 41 high and 41 low responders to hypoxia according to the median value of the hypoxic ventilatory response to hypoxia at exercise (HVRe > or < 0.84 L/min/kg) derived from the hypoxic exercise test (inspired fraction of O2: 0.115, exercise intensity of 30% of maximal aerobic power), as previously described.

The hypoxic exercise test consists in 4 successive phases of 3 to 4 minutes each with the following sequence: rest in normoxia (RN), rest in hypoxia (RH), exercise in hypoxia (EH) and exercise in normoxia (EN). Minute ventilation ( E, L.min-1) is measured through a metabograph (Vmax Encore, SensorMedics, Yorba Linda, CA). Pulse O2 saturation (SpO2, %) is measured by transcutaneous oximetry (Nellcor N-595, Nellcor, Pleasanton, CA) on a pre-warmed ear lobe. End tidal PCO2 (PETCO2) is measured by infrared thermopile (Vmax Encore, SensorMedics, Yorba Linda, CA). During the whole test, VE, SpO2 and PETCO2 were recorded breath-by-breath. Continuous blood pressure is measured by a Finapres system. Data are transferred to a computer for further spectrum analysis. A Fast Fourier Transform (FFT) is then applied to the ventilation signal in sequences of 128 points in each phase of the test. This method will allow us to detect the presence of peaks in the frequency domain of the ventilation signal. Two main parameters are derived from the FFT: the frequency in hertz (or period in seconds) of the larger peak and its power estimated as the area under the peak at ± 0.02 Hz around the peak (in L2.s-2).

The main study will be designed in order to unravel the mechanisms and role of these oscillations in ventilation. An overall population of 90 healthy subjects and 30 patients will be included in the study.

Step 1. Effect of exercise intensity.

Step 2. Effect of altitude level.

Step 3. Effect of the stimulation of central chemoreceptors by acetazolamide.

Step 4. Effect of inhibiting the peripheral chemoreceptors by hyperoxia.

Step 5. Effect of inhibiting the peripheral chemoreceptors by hyperoxia and stimulating the central chemoreceptors by hypercapnia.

Step 6. Evaluating the presence of these oscillations in patients with sleep apneas.

Step 7. Evaluating the presence of these oscillations in patients with cardiac failure.

ELIGIBILITY:
Inclusion Criteria:

* depending on the group: see definition of groups

Exclusion Criteria:

* BMI > 30
* history of severe cardiac arrhythmia
* pulmonary hypertension
* history of coronary disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects Patients with obstructive sleep apneas Patients with cardiac failure
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-06 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Periodic pattern of ventilation | The measure is made at the end of the 6-min exercise period, only once in each condition (normoxia, hypoxia, hyperoxia, hypercapnia),
  Presence of oscillation in the ventilation signal

SECONDARY OUTCOMES:
Oscillations in heart rate | The measure is made at the end of the 6-min exercise period, only once in each condition (normoxia, hypoxia, hyperoxia, hypercapnia)
  Presence of oscillations in the beat-by-beat ECG signal with a specific peak in the frequency spectrum
Oscillations in arterial blood pressure | The measure is made at the end of the 6-min exercise period, only once in each condition (normoxia, hypoxia, hyperoxia, hypercapnia)
  Presence of oscillations in the systolic/diastolic value of instant arterial blood pressure, measured non-invasively.

CONTACTS AND LOCATIONS:
Locations (1):
- Physiology Department, Bobigny, France

REFERENCES:
- [Background] Richalet JP, Larmignat P, Poitrine E, Letournel M, Canoui-Poitrine F. Physiological risk factors for severe high-altitude illness: a prospective cohort study. Am J Respir Crit Care Med. 2012 Jan 15;185(2):192-8. doi: 10.1164/rccm.201108-1396OC. Epub 2011 Oct 27. PMID 22071330
- [Derived] Hermand E, Pichon A, Lhuissier FJ, Richalet JP. Low-frequency ventilatory oscillations in hypoxia are a major contributor to the low-frequency component of heart rate variability. Eur J Appl Physiol. 2019 Aug;119(8):1769-1777. doi: 10.1007/s00421-019-04166-x. Epub 2019 Jun 1. PMID 31154522
- [Derived] Hermand E, Lhuissier FJ, Richalet JP. Effect of dead space on breathing stability at exercise in hypoxia. Respir Physiol Neurobiol. 2017 Dec;246:26-32. doi: 10.1016/j.resp.2017.07.008. Epub 2017 Jul 29. PMID 28760461